CLINICAL TRIAL: NCT03879044
Title: Transcranial Direct Current Stimulation Therapy for Sleepiness Related to Shift Work Disorder (tDCS-SWORD)
Acronym: tDCS-SWORD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding stopped
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ulysses Magalang MD, Professor of Medicine and Neuroscience Director, Sleep Medicine Program, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018H0139
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Shift-Work Sleep Disorder
Keywords: Transcranial Direct Current Stimulation
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This is a preliminary single-arm study. The study will last up to 6 weeks including the screening period. Subjects will receive active tDCS for 30 minutes before their scheduled work hours at least 3x/week for two consecutive weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Transcranial Direct Current Stimulation (Experimental): Active tDCS for 30 minutes before their scheduled work hours at least 3x/week for two consecutive weeks.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — tDCS is a form of noninvasive, painless, brain stimulation that uses a mild direct electrical current passed between electrodes on the scalp to modify neuronal membrane resting potential in a polarity dependent manner, elevating or lowering neuron excitability in a region.
  Other Names: tDCS

SUMMARY:
1. To determine the effects of tDCS on subjective measures of sleepiness in night-shift workers with shift work disorder.
2. To determine the effects of transcranial direct current stimulation (tDCS) on vigilance in night-shift workers with shift work disorder.

DETAILED DESCRIPTION:
This is a preliminary single-arm study. The study will last up to 6 weeks including the screening period. Subjects will receive active tDCS for 30 minutes before their scheduled work hours at least 3x/week for two consecutive weeks.

Outcome measures will include: psychomotor vigilance test (PVT) and the Karolinska Sleepiness Scale (KSS)25,26 which will be obtained during the shift work.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* works 5 or more night shifts per month (each shift lasting at least 10 hours, with ≥6 hours worked between 10 pm and 8 am) with plans to maintain this schedule for the duration of the 3-week trial
* meets the criteria for Shift Work Disorder according to the International Classification of Sleep Disorders24 and evaluation of a sleep medicine provider (physician or nurse practitioner) during a screening evaluation:

  1. affirmative answers to Do you experience excessive sleepiness? (yes/no); "Do you experience difficulties with falling asleep during opportunities for sleep? (yes/no); "Is the sleep or sleepiness problem related to a work schedule where you have to work when you would normally sleep? (yes/no)"; and "Has this sleep or sleepiness problem related to your work schedule persisted for at least three months? (yes/no)
  2. based on the evaluation of the sleep medicine provider, the sleep and/or wake disturbance are not better explained by another current sleep disorder, medical or neurologic disorder, mental disorder, medication use, poor sleep hygiene, or substance abuse disorder.
* Stable medication dosage over previous 4 weeks.
* Able to understand English and give a written informed consent document.

Exclusion Criteria:

* Currently taking stimulant medications such as Modafinil, Armodafinil, Methylphenidate, or Dextroamphetamine.
* History of automobile accident due to falling asleep while driving
* Inability to understand or read English
* Self-reported Substance abuse (current)
* Excessive alcohol consumption defined as:
* More than 3 glasses of wine a day
* More than 3 beers a day
* More than 60 mL of hard liquor a day
* Presence of cardiac pacemaker or automatic implantable cardioverter-defibrillator (AICD).
* Pregnancy, lactation (will be screened with urine pregnancy test)
* Non-removable metal or tattoos around head
* Use of implantable birth control device such as Implanon
* History of frequent severe headaches
* Unstable coronary artery disease
* Uncontrolled Seizure disorder
* Uncontrolled hypertension
* Any other clinically significant condition that, in the opinion of the Investigator, might put the subject at risk of harm during the study or might adversely affect the interpretation of the study data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulysses Magalang, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcranial Direct Current Stimulation
Started | 30
Completed | 26
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: We analyzed data of participants who fully complete baseline questionnaires
  years | 31.33 (7.08)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We analyzed data of participants who fully complete baseline questionnaires
  Participants
    Female | 24
    Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: We analyzed data of participants who fully complete baseline questionnaires
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 24
    Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: We analyzed data of participants who fully complete baseline questionnaires
  Participants
    American Indian or Alaska Native | 0
    Asian | 2
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 4
    White | 18
    More than one race | 2
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: We analyzed data of participants who fully complete baseline questionnaires
  Participants
    United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Psychomotor Vigilance Test
Description: Objective measure of sleepiness. Scale ranges between each individual, with the reciprocal of the reaction time being reported.
Time Frame: 3 minutes
Population: Objective sleepiness based on Psychomotor Vigilance Test could not be analyzed and reported in the table data as we were unable to collect data from enrolled patients.
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 0

2. Primary Outcome: Karolinska Sleepiness Scale
Description: Subjective measure of sleepiness. Scale ranges from 1-9, with total score being reported.
Time Frame: 5 minutes
Population: Subjective sleepiness based on Karolinska Sleepiness Scale instrument could not be analyzed and reported in the table data as we were unable to collect data from enrolled patients.
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 0

3. Secondary Outcome: Epworth Sleepiness Scale
Description: Subjective measure of sleepiness. The scale ranges from 0-24, with the total score being reported.
Time Frame: 5 minutes
Population: Subjective sleepiness based on Epworth Sleepiness Scale instrument could not be analyzed and reported in the table data as we were unable to collect data from enrolled patients.
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed through study completion (6 weeks for each participant).
Description: No adverse events were observed or reported during the study.
Arm/Group | Transcranial Direct Current Stimulation
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

LIMITATIONS AND CAVEATS:
Outcome measurements and adverse events were not analyzed and reported as the study was terminated due to funding stopped

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT03879044/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT03879044/ICF_001.pdf